CLINICAL TRIAL: NCT00454272
Title: Comparison of Teicoplanin and Vancomycin in Initial Empirical Antibiotic Regimen for Febrile Neutropenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M000507_6004
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Infection; Febrile Neutropenia
Keywords: febrile; neutropenia; cancer; Gram positive infection
MeSH Terms: conditions — Infections; Febrile Neutropenia; Fever; Neutropenia; Neoplasms | interventions — Teicoplanin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, Vancomycin (Active Comparator): Vancomycin
  Interventions: Drug: Vancomycin
- 2, Teicoplanin (Active Comparator): Teicoplanin
  Interventions: Drug: Teicoplanin

INTERVENTIONS:
Drug: Teicoplanin
  Arms: 2, Teicoplanin
Drug: Vancomycin
  Arms: 1, Vancomycin

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of Teicoplanin versus Vancomycin as part of the initial antibiotic regimen in the therapy of patients with fever and neutropenia .

ELIGIBILITY:
Inclusion Criteria:

* Will initiate study drug treatment in the hospital;
* Has a life expectancy exc. 1 month.Is male or a non-pregnant, non-lactating female, who is post-menopausal, surgically sterilized; or has been using one or more birth control methods for at least two months prior to study entry.
* Effective contraception must continue for at least 30 days after treatment discontinuation;

Exclusion Criteria:

* Has a history of suspected or documented Type I hypersensitivity reaction (e.g. anaphylactic or anaphylactoid shock, respiratory distress from bronchospasm or rash) to glycopeptides (vancomycin or teicoplanin), aminoglycosides, b-lactams or cephalosporins
* Has renal dysfunction requiring dialysis ;
* Has neutropenia associated with a syndrome that is not generally thought to be associated with a high risk of bacterial infection (e.g., chronic benign neutropenia);
* Is in blast crisis of chronic myeloid leukemia;
* Has a known underlying immunocompromising disease likely to interfere with the evaluation of therapeutic response, such as infection with human immunodeficiency virus (HIV) ;
* Had isolation and identification of a specific pathogen suspected to be responsible for fever ;Has documented colonization with vancomycin-resistant Enterococcus faecium or with Enterococcus faecalis
* Had received more than one dose of a systemic (whether oral or parenteral) antibiotic within 3 calendar days preceding the initial therapy for this episode of fever;
* Has received oral vancomycin for prophylaxis of Gram-positive infection;
* Requires addition of anti-viral, anti-anaerobic or anti-fungal coverage at the same time as study medication; however, antiviral or antifungal prophylaxis is allowed, provided that it is not started at the same time than study medication.
* Has suspected, invasive fungal disease (e.g. image of necrotic pneumonia), peri-rectal infection, liver abscess, or necrotizing enterocolitis (typhlitis).
* Had a negative serum or urine laboratory pregnancy test (for all women except those post-menopausal or surgically sterilized).
* The patient has one of the following:Leukemia, lymphoma, Hodgkin's disease, solid tumors or who had undergone bone marrow transplantation (for any reason)
* Had neutropenia at the time of initiation of initial empiric antibiotic therapy, defined as <500 neutrophils/mm3 of blood; or if ³500 but <1,000 neutrophils/mm3 and expected to fall below 500 neutrophils/mm3 within 48 hours.
* Has at least one of the following conditions:
* clinically obvious, serious catheter-related infections. For a patient with documented catheter-related infection due to an organism other than coagulase negative staphylococci, the catheter has been removed within 24 hours of identification (removal over a guidewire is permitted).
* Intensive chemotherapy that produces substantial mucosal damage (i.e., high-dose cytarabine (> 1 g/m2/day, which increases the risk for penicillin resistant streptococcal infections, particularly those due to viridans streptococci);
* prophylaxis with quinolones before the onset of the febrile episode; known colonization with pneumococci that are resistant to penicillin and -cephalosporins or methicillin-resistant S. aureus; a blood culture positive for gram-positive bacteria before final identification and susceptibility

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter will be the Response | 4 to 6 days after study drug discontinuation.

SECONDARY OUTCOMES:
Safety will be assessed for all randomized patients who received at least one dose | 1 month after the last dose of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi aventis administrative office, Istanbul, Turkey (Türkiye)